CLINICAL TRIAL: NCT02747095
Title: Clinical Investigation Plan for IQon Spectral CT at Utrecht Medical Center (UMC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Healthcare (Industry)
Collaborators: UMC Utrecht (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DHF246925
Record Dates: First submitted 2016-02-15; First posted 2016-04-21 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Artery; Deformity; Coronary (Acquired)
Keywords: CT; Spectral Images
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Spectral CT image (Experimental): Interventions: IQon Spectral CT
  Interventions: Device: IQon Spectral CT

INTERVENTIONS:
Device: IQon Spectral CT — Using IQon Spectral CT, Assess the added diagnostic value and impact on workflow of spectral images

SUMMARY:
The CT examination on IQon Spectral CT would be a standard of care CT performed as per the clinical indication. The conventional CT images generated by the scanner will be used for clinical purposes as routinely practiced. And therefore, the primary study aim is to assess the impact of IQon Spectral CT scanner and applications on the clinical workflow of the site as well as the diagnostic confidence levels of the physicians reading the CT cases.

In addition to the aim mentioned above, the investigators would like to develop recommendations for the clinical application of the spectral images in routine use. Such recommendations could include optimization of scanning protocols, optimization of reconstruction parameters; evaluate the utility of iodine maps and other supported materials.

DETAILED DESCRIPTION:
The study aim is to assess the added diagnostic value and impact on workflow of Philips IQon Spectral Computed Tomography.

The IQon Spectral CT generates two result types:

* Conventional CT images which are equivalent to images produced by the commercially available Brilliance iCT scanner
* Spectral CT images which are unique to this product.

The CT examination would be a standard of care CT performed as per the clinical indication.

In addition to the aim mentioned above, the investigators would like to develop recommendations for the clinical application of the spectral images in routine use. Such recommendations could include optimization of scanning parameters, optimization of reconstruction parameters to utilize the capabilities of the IQon system etc.

The clinical system includes:

* The IQon Spectral CT scanner
* Spectral Diagnostic suite (Philips IntelliSpace Portal): includes 5 applications. Spectral Enhanced CT Viewer, Spectral Enhanced Advanced Analysis, Spectral Enhanced Comprehensive Cardiac Analysis, Spectral Enhanced Tumor Tracking, spectral magic glass on PACS.

The testing will be conducted under this project plan. This is a single center research study that is expected to be conducted over a one year period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects clinically indicated to have a CT scan as part of their routine, standard medical care. Subjects must be capable of providing informed consent for the retrospective use and analysis of the IQon Spectral CT data for the research study.

Exclusion Criteria:

* Subjects that are not clinically indicated to have a CT scan as part of their routine, standard medical care. Subjects that are not capable of providing informed consent for the retrospective use and analysis of the IQon Spectral CT data for the research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 980 (Actual)
Dates: Start 2016-01; Primary Completion 2017-04-28 (Actual); Study Completion 2017-04-28 (Actual)

PRIMARY OUTCOMES:
Degree of improvement in specificity (measures the proportion of negatives that are correctly identified) of spectral coronary CTA for detection of coronary stenoses in need of treatment over conventional coronary CTA | One Year

SECONDARY OUTCOMES:
Change in sensitivity (measures the proportion of positives that are correctly identified) of SDCT versus conventional CT scanning for characterizing pulmonary nodules. | One Year
Change in specificity (measures the proportion of negatives that are correctly identified) of SDCT versus conventional CT scanning for characterizing pulmonary nodules. | One Year
Change in sensitivity (measures the proportion of positives that are correctly identified) of SDCT versus conventional CT scanning or characterizing carotid atherosclerotic plaque components | One Year
Change in specificity (measures the proportion of negatives that are correctly identified) of SDCT versus conventional CT scanning or characterizing carotid atherosclerotic plaque components | One Year

CONTACTS AND LOCATIONS:
Overall Officials: Tim Leiner, Principal Investigator — Utrect Medical Center
Locations (1):
- Utrecht Medical Center, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No